CLINICAL TRIAL: NCT05025722
Title: An Evaluation of Pseudoxanthoma Elasticum (PXE) Natural History Biomarkers in PXE Individuals and Their Biological Non-PXE Siblings
Brief Title: Pseudoxanthoma Elasticum (PXE) Natural History Biomarkers in PXE Individuals and Their Biological Non-PXE Siblings
Status: Completed | Type: Observational
Sponsor: Daiichi Sankyo (Industry)
Collaborators: PXE International (Other); Thomas Jefferson University (Other)
Responsible Party: Sponsor
Other Study IDs: DS1211-A-U104
Record Dates: First submitted 2021-07-30; First posted 2021-08-27 (Actual); Last update posted 2022-09-06 (Actual); Status verified 2022-09

CONDITIONS: Pseudoxanthoma Elasticum
Keywords: Pseudoxanthoma Elasticum; Bone turnover biomarkers; Tissue mineralization biomarkers
MeSH Terms: conditions — Pseudoxanthoma Elasticum

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Confirmed PXE participants: Participants who have index PXE/proband with established PXE and ABCC6 mutations identified.
  Interventions: Other: Non Interventional
- PXE carrier participants: Participants who are biological siblings of the PXE index case and confirmed as PXE carrier.
  Interventions: Other: Non Interventional
- Non-PXE normal participants: Participants who are biological siblings of PXE index case and confirmed as non-PXE normal.
  Interventions: Other: Non Interventional

INTERVENTIONS:
Other: Non Interventional — This is an observational study.

SUMMARY:
This PXE biomarker study aims to characterize the levels of inorganic pyrophosphate (PPi), pyridoxal 5´-phosphate (PLP), and other biomarkers relevant to PXE and ectopic calcification in both PXE patients and their biological siblings who are PXE carriers or normal non-PXE individuals.

DETAILED DESCRIPTION:
This non-interventional PXE study is designed to assess differences in circulation levels of selective biomarkers related to PXE and tissue-nonspecific alkaline phosphatase (TNAP) inhibition, between PXE patients, PXE carriers, and non-PXE normal individuals.

ELIGIBILITY:
Inclusion Criteria:

* Male or female participants aged 18 to 75 years
* Participants (approximately 1 carrier and 1 normal to match proband)

  * Confirmed PXE participants: index PXE/proband with established PXE and ABCC6 mutations identified
  * PXE carrier participants: biological sibling of the PXE index case and confirmed as PXE carrier
  * Non-PXE normal participants: biological sibling of PXE index case and confirmed as non-PXE normal

Exclusion Criteria:

* Unconfirmed ABCC6 mutation status
* Use of bisphosphonate in the preceding 12 months and during the study
* Use of Vitamin B6 and/or Vitamin D supplement in the preceding 1 month and during the study (if the total Vitamin B6 supplementation is >5 mg/day)
* Recent initiation or dose change of Vitamin D and/or multivitamin supplement in the preceding 1 month and during the study
* Bone fracture within 3 months prior to Screening or active bone disease (excluding osteopenia or osteoporosis)
* History of hyperparathyroidism
* History of moderate to severe renal impairment
* History of hypophosphatasia
* Known history of uncorrected abnormality in calcium (Ca), phosphate, alkaline phosphatase (ALP) or parathyroid hormone
* Other significant condition (medical, psychiatric, social, or medication) that, in the judgment of the Investigator, would prevent full participation or would be inappropriate for the study

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: PXE probands with identified ABCC6 mutations and non-PXE biological siblings will be invited for study participation.
Sampling Method: Non-Probability Sample
Enrollment: 48 (Actual)
Dates: Start 2021-08-30 (Actual); Primary Completion 2022-08-11 (Actual); Study Completion 2022-08-11 (Actual)

PRIMARY OUTCOMES:
Mean Plasma Levels of Inorganic Pyrophosphate (PPi) | Study visit (0 up to 2 hours)
  PPi will be assessed by study group and by timepoint where applicable.
Mean Plasma Levels of Pyridoxal 5´-Phosphate (PLP) | Study visit (0 up to 2 hours)
  PLP will be assessed by study group and by timepoint where applicable.
Mean Serum Enzyme Activity Levels of Alkaline Phosphatase (ALP) | Study visit (0 up to 2 hours)
  ALP will be measured using the standard clinical chemistry assays, by study group and by timepoint where applicable.
Mean Serum Enzyme Activity Levels of Bone-specific Alkaline Phosphatase (BSAP) | Study visit (0 hours)
  BSAP will be measured using the standard clinical chemistry assays, by study group and by timepoint where applicable.

SECONDARY OUTCOMES:
Percent Change from Baseline in Plasma Levels of PPi and PLP, by Sex | Study visit (0 to 2 hours)
  Blood samples will be assessed by sex group.
Percent Change from Baseline in Serum Enzyme Activity of ALP, by Sex | Study visit (0 to 2 hours)
  Blood samples will be assessed by sex group.
Percent Change from Baseline and Variability in Plasma Levels of PPi and PLP | Study visit (0 to 2 hours)
  Variability of PPi and PLP will be assessed.
Percent Change from Baseline and Variability in Serum Enzyme Activity of ALP | Study visit (0 to 2 hours)
  Variability of ALP will be assessed.

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Leader, Study Director — Daiichi Sankyo
Locations (1):
- Thomas Jefferson University, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No